CLINICAL TRIAL: NCT07102654
Title: Comparison Between Digital Nerve Microanastomosis and Traction Neurectomy in Post-Digital Amputation Pain: A Prospective Study
Brief Title: Comparison Between Digital Nerve Microanastomosis and Traction Neurectomy in Post-Digital Amputation Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2026-13097
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-07

CONDITIONS: Amputation Stump; Amputation Neuroma; Amputation, Traumatic/Surgery; Amputation, Surgical
Keywords: microanastomosis; traction neurectomy; digital amputation; digital nerve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to assess the post-operative pain in adults with digital amputation following two different surgical interventions: microanastomosis of digital nerves or traction neurectomy. The main questions it aims to answer are:

* Which surgical intervention results in less post-operative pain?
* Which surgical intervention leads to fewer symptoms after six months?
* Which surgical intervention is associated with fewest post-operative complications? Participants will complete a Visual Analog Scale (VAS) to assess the pain and the Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) to evaluate the disabilities.

The researchers will assess post-operative complications during follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who have undergone a traumatic digital amputation
* Patients treated with one of the two following techniques: microanastomosis of digital nerves or traction neurectomy
* Postoperative follow-up of at least 6 months

Exclusion Criteria:

* Patients treated with a surgical intervention other than microanastomosis of digital nerves or traction neurectomy for digital amputation
* Non-traumatic amputations (e.g., cancer or infection)
* Follow-up of less than 6 months
* Patients with pre-existing peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals presenting at the Centre Hospitalier de l'Université de Montréal for a digital amputation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Measured by Visual Analog Scale in Adult Patients Following Digital Amputation | 1 week, 4 weeks and 6 months
  The primary objective of this study is to compare the level of postoperative pain associated with two surgical techniques: microanastomosis of digital nerves and traction neurectomy. Pain will be measured using the visual analog scale at one week, four weeks, and six months following the procedure. The visual analog scale ranges from 0 ( no pain) to 10 (worst imaginable pain).
Postoperative Symptoms Measured by the Disabilities of the Arm, Shoulder and Hand Questionnaire in Adult Patients Following Digital Amputation | 6 months
  The secondary objective of this study is to compare the level of postoperative symptoms associated with two surgical techniques: microanastomosis of digital nerves and traction neurectomy. The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will assess disability and hand-related symptoms at 6 months. The score ranges from 0 (no disability) to 100 (most severe disability)

SECONDARY OUTCOMES:
Complication Rate of Microanastomosis of Digital Nerves and Traction Neurectomy in Adult Patients Following Digital Amputation | 1 week, 4 weeks, 6 months
  The tertiary objective of this study is to determine the incidence of postoperative complications for both microanastomosis of digital nerves and traction neurectomy.